CLINICAL TRIAL: NCT01347489
Title: Cronic Pressure Wounds and Relation With Gender
Acronym: preswound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: SB Istanbul Education and Research Hospital (Other)
Responsible Party: Erhan Aysan, Assoc. Prof.
Other Study IDs: 3-Aysan
Record Dates: First submitted 2011-05-03; First posted 2011-05-04 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2010-11

CONDITIONS: Wound
Keywords: gender
MeSH Terms: conditions — Wounds and Injuries; Coitus

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There is no exact scientfic data about gender relationship with cronic pressure wounds (CPW). This research is aimed first to reveal gender relationship with CPW and aimed secondarily to reveal the gender related couse(es).

DETAILED DESCRIPTION:
There is no exact scientific data about gender relationship with cronic pressure wounds (CPW). Researches about this subject is generally related to prevention and management of the process. But gender difference is not exactly researched in the literature. This research is aimed first to reveal gender relationship with CPW and aimed secondarily to reveal the gender related couse(es).

ELIGIBILITY:
Inclusion Criteria:

* Cronic pressure wound patients

Exclusion Criteria:

* Operated cronic pressure wounds

Ages: 17 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cronic pressure wound patients
Sampling Method: Non-Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-06 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: erhan aysan, Assoc. Prof., Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)